CLINICAL TRIAL: NCT03847259
Title: Mechanical Posture Changes in Adolescent Female at Public Schools Compared to International Schools
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, Lecturer of biomechanics, Cairo University
Other Study IDs: MPCAF
Record Dates: First submitted 2019-01-10; First posted 2019-02-20 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A(public school): it will be consists of 200 adolescent female from public schools, their age will be ranged from 13 to 17 years, initiated menstrual cycle and BMI more than 20.mechanical posture changes will be evaluated by Posture screen mobile. back pain and life style will be evaluated by (BackPEI) questionnaire.
  pain will be evaluated by VISUAL ANALOG SCALE(VAS) .stress will be evaluated by Depression Anxiety Stress Scales-21(DASS-21).
  Interventions: Diagnostic Test: mechanical posture changes
- B(international school): it will be consists of 200 adolescent female from international schools their age will be ranged from 13 to 17 years, initiated menstrual cycle and BMI more than 20.mechanical posture changes will be evaluated by Posture screen mobile. back pain and life style will be evaluated by (BackPEI) questionnaire .pain will be evaluated by VISUAL ANALOG SCALE (VAS).stress will be evaluated by Depression Anxiety Stress Scales-21(DASS-21).
  Interventions: Diagnostic Test: mechanical posture changes

INTERVENTIONS:
Diagnostic Test: mechanical posture changes — evaluated by Posture screen mobile, (BackPEI) questionnaire , VISUAL ANALOG SCALE (VAS), Depression Anxiety Stress Scales-21(DASS-21).

SUMMARY:
The aim of this study is to determine different mechanical posture changes in adolescent females at public schools compared to international schools.

DETAILED DESCRIPTION:
Two hundred adolescent female subjects at public schools and in this study. All subjects will be recruited from different schools. 1-Group A: it will be consists of 200 adolescent female from public schools, will be evaluated by Posture screen mobile, (BackPEI) questionnaire , VISUAL ANALOG SCALE (VAS)and Depression Anxiety Stress Scales-21(DASS-21).

2- Group B: it will be consists of 200 adolescent female from international schools, will be evaluated by Posture screen mobile, (BackPEI) questionnaire , VISUAL ANALOG SCALE (VAS) and Depression Anxiety Stress Scales-21(DASS-21).

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent female at schools.
2. Their age will be ranged from 13 to 17 years.
3. BMI more than 20.
4. Initiated menstrual cycle.

Exclusion Criteria:

1. Asthma and chronic respiratory disease.
2. History of upper and lower limb injury.
3. Under weight subjects.
4. Females with congenital spinal deformities.
5. Diabetes, cardiopulmonary diseases and any physical impairment that prevent following the study program.

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — both boys and g( da Rosa et al., 2017). They found that girls had poor posture due to the way they carried their school supplies (da Rosa et al., 2017).irls presented a constant frequency in back pain and poor sitting posture, but girls presented higher prevalence along
Study Population: Adolescent female at schools.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
posture deviations | up to 6months
  Lateral shift from the midline and tilting through frontal and lateral views.

SECONDARY OUTCOMES:
weight | up to 6months
  Anthropometric measurement measure by kilogram (kg).
height | up to 6months
  Anthropometric measurement measure by centimeter (cm).
body mass index (BMI). | up to 6 months
  calculated by dividing weight (in kilograms) by your height (in metres squared). kg/m2
Back Pain and Body Posture Evaluation Instrument (BackPEI) questionnaire | up to 6months
  Back Pain and Body Posture Evaluation Instrument .The BackPEI questionnaire consists of 21 closed questions, which address the occurrence, frequency and intensity of pain, as well as questions on demographic (age, gender) and behavioral factors (level of exercise, competitive or non-competitive practice of exercise, daily hours watching television and using the computer, number of daily hours of sleep, reading and/or studying in bed, and postures in activities of daily living.
Visual analogue scale | up to 6months
  Numerical pain rating scale (minimum score 0 and maximum score 10) ,Instruct the patient to choose a number from 0 to 10 that best describes their current pain. 0 would mean "no pain" and 10 would mean "worst possible pain.
Depression Anxiety Stress Scales-21(DASS-21) | up to 6months
  Was developed to provide a self-report measure of anxiety, depression and stress signals. During the development process.Questionnaire consists of 21 questions,seven questions for depression ,seven for anxiety and seven for stress assessment.The responses are given on a 4-point Likert scale, ranging from zero if "I strongly disagree" to 3 if "I totally agree". Overall scores for the three constructs are calculated as the sum of scores for the relevant seven items multiplied by two. Ranges of scores correspond to levels of symptoms, ranging from "normal" to "extremely serious

CONTACTS AND LOCATIONS:
Overall Officials: fahema me okeel, phD, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided